CLINICAL TRIAL: NCT01909180
Title: Clinical Evaluation for GE CT System
Brief Title: Clinical Evaluation for General Electric (GE) CT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 106-2011-GES-0003
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: CT Scanners X Ray

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cardiac (Experimental): Revolution CT Cardiac Imaging Scan
  Interventions: Device: Revolution CT Scanner
- Body/Extremity (Experimental): Revolution CT Body and/or Extremity Imaging Scan
  Interventions: Device: Revolution CT Scanner
- Neuro (Experimental): Revolution CT Brain and Spinal Cord Imaging Scan
  Interventions: Device: Revolution CT Scanner

INTERVENTIONS:
Device: Revolution CT Scanner — These scans would be considered "standard of care" but, because the subjects are scanned on an uncleared device they are investigational.

SUMMARY:
An external evaluation to obtain clinical data to create sample clinical images.

The data will also be used for product and technology development, marketing materials, and inclusion in publications.

DETAILED DESCRIPTION:
The image data were assessed using a Likert scale for image quality sufficient for diagnostic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily signed the Informed Consent Form (ICF).
* Male subjects 18 years of age or older.
* Female subjects 18 years of age or older. Females between 18 and 60 years of age must be non-lactating and non-pregnant as confirmed by negative urine pregnancy test., unless they had surgery resulting in sterilization or are post-menopausal according to the medical history.

Exclusion Criteria:

* • Subjects previously enrolled in this Evaluation.

  * Subjects who are not able or not willing to give written Informed Consent.
  * For IV contrast-enhanced CT exams, anyone with known or suspected allergy to iodinated contrast agents or a history of multiple allergies or asthma.
  * For IV contrast-enhanced CT exams, per the institution's guidelines on risk stratification and prophylaxis for Contrast Induced Neuropathy, subjects will be pre-screened via medical history review by qualified medical personnel for suspected renal function impairment and high risk subjects will undergo a serum creatinine lab test. Any subject with proven renal insufficiency will be excluded.
  * Known pregnancy and nursing (lactating) females.
  * Any subject with urgent medical condition requiring acute care.
  * Any conditions that, in the opinion of the Investigator, would interfere with the evaluation of the results or constitute a health hazard for the subject.
  * Subjects who do not agree to allow GEHC personnel to be present during the scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Curry, MD, Principal Investigator — Baptist South Hospital
Locations (1):
- Baptist South Florida Hospital, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Scan: This is a single arm clinical trial.
  Standard of care scan
  Investigational Scan
Period: Overall Study
Arm/Group | Standard of Care Scan
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Standard of Care Scan
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Image Quality
Description: Image quality assessment on a 5 point Likert Scale:
  5= Diagnostic- Excellent Image Quality 4= Diagnostic- Good Image Quality 3= Diagnostic-Acceptable Image Quality 2= Sub-Optimal Diagnostic with limited additional clinical information
  1= Non-Diagnostic
Time Frame: 24 hours
Population: All cases were sufficient and had acceptable, good or excellent image quality
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Scan Images
Groups:
- Cardiac: Subjects who received a cardiac CT scan
- Body/ Extremity: Subject receiving a Revolution CT scan of the body or extremities
- Neuro: Subjects receiving Revolution CT Scans of Brain or Spinal Cord
Arm/Group | Cardiac | Body/ Extremity | Neuro
Number analyzed (Participants) | 19 | 20 | 10
Number analyzed (Scan Images) | 57 | 60 | 30
units on a scale | 4.53 (0.68) | 4.44 (0.67) | 4.63 (0.61)

ADVERSE EVENTS:
Arm/Group | Standard of Care Scan
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 1/49
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Scan (N=49)
Vomitting (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No